CLINICAL TRIAL: NCT00489437
Title: Improving the Diagnosis of Heparin-Induced Thrombocytopenia: Utility of the 4T's Score and Evaluation of New Rapid Assays
Brief Title: Heparin-Induced Thrombocytopenia Score Card Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HHS06-451
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Heparin-Induced Thrombocytopenia
Keywords: diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ID-PaGIA Heparin/PF4 antibody test — All patients have a 4T's Score completed, a same-day PaGIA performed and a Serotonin Release Assay performed.
Procedure: Clinical Prediction Score-HIT Score Card — 1. clinical prediction rule
  2. rapid immunoassay

SUMMARY:
Main Research Question:

Can two new types of test, one called the 4T's score and the other called a rapid assay, help doctors correctly identify which patients are unlikely to have heparin-induced thrombocytopenia (HIT)?

HIT is a severe allergic reaction to the blood thinner heparin. This allergic reaction can lead to heart attacks, strokes, limb amputations, and death. Because heparin is one of the most commonly used drugs in the hospital setting, it is very important that the investigators are able to correctly identify who can safely continue to take heparin and who cannot.

It can be very difficult to diagnose HIT because it can look like many other medical conditions and the best laboratory tests for HIT are difficult to run and only available at specialized centres.

It would be very helpful if doctors had tests they could use that would tell them quickly and accurately which patients with symptoms that look like HIT really do have HIT (and require urgent treatment with another type of blood thinner) and which patients are very unlikely to have HIT (and could continue to take heparin safely). In this study, the investigators will compare the 4T's score (a scoring system that assigns "points" to the presence or absence of specific clinical features) and a rapid laboratory test with the old laboratory test to find out if one or both of these types of tests are useful for telling doctors which patients have HIT and which patients don't have HIT.

ELIGIBILITY:
Inclusion Criteria:

* Suspected heparin-induced thrombocytopenia

Exclusion Criteria:

* Unable to give consent
* Unable to provide a blood sample
* Previous entered in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2007-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a low or intermediate 4T's Score and a negative ID-PaGIA assay result who have a positive SRA. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lori-Ann Linkins, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Linkins LA, Bates SM, Lee AY, Heddle NM, Wang G, Warkentin TE. Combination of 4Ts score and PF4/H-PaGIA for diagnosis and management of heparin-induced thrombocytopenia: prospective cohort study. Blood. 2015 Jul 30;126(5):597-603. doi: 10.1182/blood-2014-12-618165. Epub 2015 Apr 29. PMID 25926600